CLINICAL TRIAL: NCT05569135
Title: Debridement and Laser Ablation Versus Debridement Alone in Pilonidal Disease: Retrospective Analysis of Mid-term Outcome
Brief Title: Debridement and Laser Ablation Versus Debridement Alone in Pilonidal Disease
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: E-10840098-772.02-2926
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Pilonidal Disease
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Debridement only: Debridement of the pilonidal cyst through pits was performed in this group. After the removal of hair and necrotic tissues through pits, the surgical site was covered with a simple gauze dressing for 1 day. Patients were allowed to return to work and sit freely on the day of surgery.
- Debridiment with laser ablation: This group underwent the same procedure as the debridement group. After the removal of hair and necrotic tissues through pits, a diode laser at 1470 wavelength was inserted and the pilonidal cavity was ablated in a continuous fashion. The surgical site was covered with a simple gauze dressing for 1 day. Patients were allowed to return to work and sit freely on the day of surgery.
  Interventions: Device: Laser ablation

INTERVENTIONS:
Device: Laser ablation — A diode-laser that has been reported to be safe and effective in several treatments including pilonidal disease, anal fistula, hemorrhoids, and vascular ablation was used to obtain shrinkage of pilonidal cyst
  Groups: Debridiment with laser ablation

SUMMARY:
This study aims to investigate the effect of laser ablation (LA) in minimally invasive management of pilonidal disease (PD).

Data of the patients with PD who were eligible for simple debridement have been prospectively collected since March 2018, when laser ablation treatment came into use in our institution. Laser ablation treatment was offered to all eligible patients. All the patients underwent debridement (removal of hair and/or necrotic tissues through pits using a clamp/curette/brush) of PD; LA was added to the procedure in patients who were willing to have LA. The surgical outcome of two procedures was compared. The primary outcome measure was recurrence at 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Class III, IV, and V pilonidal disease according to Tezel Navicular Area Classification
* Patients who underwent debridement for pilonidal disease

Exclusion Criteria:

* Patients with acute abscess (Tezel Class II)
* Antibiotic use within 4 weeks before surgery
* Patients lost to follow-up at 3,7 and 30 days; 6, 12 and 36 months

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Female and males older than 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
disease recurrence at 36 months | 36 months
  Any ongoing or recurrent sypmtoms were recorded

SECONDARY OUTCOMES:
Complications after the procedure | 1 month
  Safety of the procedure
Incidence of adverse events | 1 month
  Safety of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Naciye Cigdem Arslan, MD, Principal Investigator — Medipol University
Locations (1):
- Medipol Bahcelievler Hospital, Istanbul, Other (Non U.s.), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tezel E. A new classification according to navicular area concept for sacrococcygeal pilonidal disease. Colorectal Dis. 2007 Jul;9(6):575-6. doi: 10.1111/j.1463-1318.2007.01236.x. No abstract available. PMID 17573759